CLINICAL TRIAL: NCT03138798
Title: Dental Support Device in the Second Stage of Labor at a Major Tertiary Care Center; A Randomized Controlled Trial
Brief Title: Dental Support Device in the Second Stage of Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Angela Bianco (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor-Investigator, Angela Bianco, Director, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 16-2121
Record Dates: First submitted 2017-04-06; First posted 2017-05-03 (Actual); Results first posted 2018-12-11 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-11

CONDITIONS: Labor
Keywords: Labor; Second stage; Dental device
MeSH Terms: interventions — Occlusal Splints

STUDY DESIGN:
Intervention Model Description: Patients will give consent in the first stage of labor. Randomization will then be performed using sealed envelopes at the time of pushing in the second stage of labor. Duration of the second stage and time spent pushing will be recorded for both groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Laboraide TM dental support device (Experimental): Receive Laboraide
  Interventions: Device: Laboraide TM dental support device
- Control Group (No Intervention): Patients will give consent in the first stage of labor. Subsequently, randomization will be performed using sealed envelopes opened at the time of pushing in the second stage of labor. Women assigned to Group B will not receive a Laboraide TM dental support device. Duration of the second stage and time spent pushing will be recorded. Obstetric management will not be altered by group assignment.

INTERVENTIONS:
Device: Laboraide TM dental support device — Patients will give consent in the first stage of labor. Subsequently a randomization will be performed using sealed envelopes opened at the time of pushing in the second stage of labor. Women assigned to Group A will received a sealed Laboraide TM package. Duration of the second stage and time spent pushing will be recorded. Obstetric management will not be altered by group assignment. Following delivery, patients assigned to Group A will complete a patient satisfaction survey.
  Other Names: Dental Device; Dental Support Device
  Arms: Laboraide TM dental support device

SUMMARY:
Obstetric practices now allow for prolonged second stage of labor to accomplish vaginal delivery. However, this practice may lead to either operative delivery (vacuum or forceps assisted delivery) or cesarean section with significant maternal/neonatal morbidity. Limited evidence suggests that dental support devices (DSD) may improve lead to shortened labor by allowing patients to push more effectively.

DETAILED DESCRIPTION:
In an effort to reduce the rate of cesarean section, obstetric practices now allow for prolonged second stage of labor to accomplish vaginal delivery. However, this practice is not without risks and may lead to either operative delivery (vacuum or forceps assisted delivery) or cesarean section with significant maternal/neonatal morbidity. Limited evidence suggests that dental support devices (DSD) may improve maternal valsalva and lead to a shortened second stage of labor by allowing them to push more effectively. Previous studies have been underpowered to find statistically significant results.

The Icahn School of Medicine at Mount Sinai has a unique and heterogeneous inner-city population of laboring mothers with marked rates of maternal obesity. The objective is to conduct a randomized controlled trial in which nulliparous patients are asked to use the LaboraideTM, a DSD designed for laboring women, while pushing with contractions in the second stage of labor.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women
* Non-anomalous fetus
* Singleton fetus
* Vertex presentation
* In the first phase of labor
* Full term gestation (>=37w0d)
* Maternal age 18-64 years

Exclusion Criteria:

* Multiparity
* History of prior uterine surgery such as cesarean section or myomectomy
* Unexplained vaginal bleeding
* Latex allergy
* Contraindication to vaginal delivery
* Pregestational or Gestational Diabetes
* Fetal growth restriction
* Fetus with suspected macrosomia
* Prematurity (<37 weeks gestational age)
* Multiple gestation
* Refusal to participate

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 348 (Actual)
Dates: Start 2017-01-06 (Actual); Primary Completion 2017-11-07 (Actual); Study Completion 2017-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Bianco, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Eric Bergh, MD, Study Director — Ichan School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Laboraide TM Dental Support Device: Laboraide TM dental support device (a commercially available dental device made of soft plastic, 3 mm in thickness, which is inserted over the lower jaw with bite plates overlying the molar teeth) and were instructed to bite down on the dental support device (DSD) while pushing.
- Control Group: no device
Period: Overall Study
Arm/Group | Laboraide TM Dental Support Device | Control Group
Started | 173 | 175
Randomized But Did Not Meet Eligibility | 6 | 4
Completed | 167 | 171
Not Completed | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Laboraide TM Dental Support Device: Laboraide TM dental support device
- Total: Total of all reporting groups
Arm/Group | Laboraide TM Dental Support Device | Control Group | Total
Number analyzed (Participants) | 167 | 171 | 338
Age, Customized [Count of Participants; unit: Participants]
  Maternal Age: 18-29 years | 58 | 56 | 114
  Maternal Age: 30-34 years | 73 | 83 | 156
  Maternal Age: 35-39 years | 32 | 27 | 59
  Maternal Age: 40+ years | 4 | 5 | 9
Age, Customized [Count of Participants; unit: Participants]
  Gestational Age at procedure: 37.0 - 38.9 weeks | 31 | 34 | 65
  Gestational Age at procedure: 39.0 - 40.9 weeks | 112 | 112 | 224
  Gestational Age at procedure: 41.0 - 41.9 weeks | 24 | 25 | 49
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 167 | 171 | 338
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 121 | 128 | 249
  African American | 8 | 7 | 15
  Asian | 10 | 14 | 24
  Hispanic | 18 | 19 | 37
  Other | 10 | 3 | 13
BMI at delivery [Count of Participants; unit: Participants] — Body Mass Index (BMI) at delivery
  Participants
    18-29 kg/m2 | 126 | 127 | 253
    30-39 kg/m2 | 35 | 43 | 78
    40+ kg/m2 | 6 | 1 | 7
Preeclampsia with severe features on Magnesium [Count of Participants; unit: Participants] | 3 | 2 | 5
Indications for Admission [Count of Participants; unit: Participants]
  Labor induction (intact membranes) | 42 | 43 | 85
  Premature rupture of membranes (PROM) | 31 | 31 | 62
  Spontaneous Labor | 94 | 97 | 191
Membrane Status [Count of Participants; unit: Participants] — Rupture of membranes (ROM) prior to admission
  Participants | 42 | 29 | 71
Meconium at ROM [Count of Participants; unit: Participants] — Meconium at Rupture of Membranes (ROM)
  Participants | 20 | 30 | 50
Cervical dilation at admission >= 6 cm [Count of Participants; unit: Participants] | 12 | 7 | 19
Number of patients on pitocin in labor [Count of Participants; unit: Participants] | 110 | 122 | 232
Epidural [Count of Participants; unit: Participants] | 148 | 154 | 302
Number anesthetic boluses administered in 2nd stage [Count of Participants; unit: Participants] — Population: Only those participants who had an epidural were included
  Participants
    number analyzed (Participants) | 148 | 154 | 302
    0 | 122 | 138 | 260
    1 | 19 | 10 | 29
    2 | 3 | 4 | 7
    3 | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Dilation Duration of Second Stage of Labor Time
Description: At the time of pushing in the second stage of labor, the time from full dilation to delivery during the second stage of labor in patients with vaginal delivery (spontaneous, vacuum, forceps included). Intention to treat analysis.
Time Frame: Up to 3 hours
Population: Only participants who delivered vaginally were included in the analysis
Measure: Median (Inter-Quartile Range); unit: minutes
Groups:
- Laboraide TM Dental Support Device: Laboraide TM dental support device (a commercially available dental device made of soft plastic, 3 mm in thickness, which is inserted over the lower jaw with bite plates overlying the molar teeth) and were instructed to bite down on the DSD while pushing.
Arm/Group | Laboraide TM Dental Support Device | Control Group
Number analyzed (Participants) | 161 | 161
minutes | 82 [40 to 122] | 90 [45 to 140]

2. Primary Outcome: Delivery Time
Description: The time from initiation of pushing until delivery during the second stage of labor. Intention to treat analysis will be performed.
Time Frame: An average of 75 minutes
Population: Only those participants who delivered vaginally were included in the analysis
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Laboraide TM Dental Support Device | Control Group
Number analyzed (Participants) | 161 | 161
minutes | 46 [23 to 80] | 53 [26 to 86]

3. Secondary Outcome: Dental Support Device Comfort and Patient Satisfaction
Description: After delivery patients assigned to the intervention group completed a comfort and satisfaction survey which consisted of three questions and given choices from strongly disagree to strongly agree
Time Frame: Post-Op Day 1
Population: Only those who participated in survey was included
Measure: Count of Participants; unit: Participants
Groups:
- Laboraide TM Support Device: Laboraide TM dental support device (a commercially available dental device made of soft plastic, 3 mm in thickness, which is inserted over the lower jaw with bite plates overlying the molar teeth) and were instructed to bite down on the DSD while pushing.
Arm/Group | Laboraide TM Support Device
Number analyzed (Participants) | 124
Participants
  Was the device comfortable: Strongly disagree | 11
  Was the device comfortable: Disagree | 15
  Was the device comfortable: Neither agree nor disagree | 15
  Was the device comfortable: Agree | 61
  Was the device comfortable: Strongly agree | 22
  Was this device helpful?: Strongly disagree | 10
  Was this device helpful?: Disagree | 12
  Was this device helpful?: Neither agree nor disagree | 27
  Was this device helpful?: Agree | 46
  Was this device helpful?: Strongly agree | 29
  Would you use the device again: Strongly disagree | 10
  Would you use the device again: Disagree | 20
  Would you use the device again: Neither agree nor disagree | 19
  Would you use the device again: Agree | 43
  Would you use the device again: Strongly agree | 32

4. Secondary Outcome: Mode of Delivery
Description: Delivery Outcomes: Mode of delivery
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Laboraide TM Dental Support Device | Control Group
Number analyzed (Participants) | 167 | 171
Participants
  Normal spontaneous vaginal delivery (NSVD) | 143 | 141
  Forcep delivery | 11 | 13
  Vacuum delivery | 7 | 7
  Cesarean section | 6 | 10

5. Secondary Outcome: Estimated Blood Loss
Description: Estimated blood loss (EBL) during delivery
Time Frame: Day 1
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Laboraide TM Dental Support Device | Control Group
Number analyzed (Participants) | 167 | 171
mL | 320 [221 to 400] | 350 [250 to 500]

6. Secondary Outcome: Number of Participants With Post-partum Hemorrhage
Description: Number of participants with post-partum hemorrhage caused by uterine atony which is a loss of tone in the uterine musculature.
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Laboraide TM Dental Support Device | Control Group
Number analyzed (Participants) | 167 | 171
Participants | 19 | 12

7. Secondary Outcome: Number of Participants With Chorioamnionitis
Description: Chorioamnionitis - an intra-amniotic infection (IAI) is an inflammation of the fetal membranes (amnion and chorion) due to a bacterial infection.
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Laboraide TM Dental Support Device | Control Group
Number analyzed (Participants) | 167 | 171
Participants | 8 | 16

8. Secondary Outcome: Neonatal Birth Weight
Description: Neonatal outcomes - birth weight
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Laboraide TM Dental Support Device | Control Group
Number analyzed (Participants) | 167 | 171
grams | 3343 (388) | 3286 (371)

9. Secondary Outcome: Neonatal Sex
Description: Neonatal outcomes - Number of male neonatal sex
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Laboraide TM Dental Support Device | Control Group
Number analyzed (Participants) | 167 | 171
Participants | 85 | 85

10. Secondary Outcome: Number of NICU Admission
Description: Neonatal outcomes: Number of neonatal intensive care unit (NICU) admissions
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Laboraide TM Dental Support Device | Control Group
Number analyzed (Participants) | 167 | 171
Participants | 17 | 14

ADVERSE EVENTS:
Time Frame: Adverse events not collected
Description: Adverse events not collected
Arm/Group | Laboraide TM Dental Support Device | Control Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-27): https://cdn.clinicaltrials.gov/large-docs/98/NCT03138798/Prot_SAP_000.pdf